CLINICAL TRIAL: NCT00070434
Title: A Phase II Feasibility Translational Research Trial of Induction Chemotherapy Followed by Concomitant Chemoradiation in Patients With Clinical T4 Rectal Cancer
Brief Title: S0304 Induct Chemo Then Chemo-RT in Pts w/Locally Advanced Adenocarcinoma of the Rectum
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000334469; U10CA032102 (NIH); S0304 (Other: SWOG)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin; Radiotherapy; Pyridoxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Irinotecan + 5-FU + Leucovorin (Experimental): Irinotecan 180mg/m2, IV for 90min on Day 1, q 2 wk x 4 cycles; 5-FU 400 mg/m2, IV bolus on Day 1, q 2 wk x 4 cycles; 5-FU 2.4 g/m2 IV for 46 hours on Day 1, q 2 wk x 4 cycles; Leucovorin 200 mg/m2 IV for 2 hours on Day 1, q 2 wk x4 cycles.
  Interventions: Drug: capecitabine; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Radiation: radiation therapy; Drug: Pyridoxine
- Irinotecan + Oxaliplatin (Experimental): Irinotecan 175mg/m2 IV for 90 minutes on Day 1, q 2wk x4 cycles; Oxaliplatin 85mg/m2 IV for 2 hours on Day 1, q 2wk x4 cycles
  Interventions: Drug: capecitabine; Drug: irinotecan hydrochloride; Drug: oxaliplatin; Radiation: radiation therapy; Drug: Pyridoxine
- Oxaliplatin + 5-FU + Leucovorin (Experimental): Oxaliplatin 85mg/m2 IV for 90 minutes on Day 1, q 2wk x4 cycles; 5-FU 400mg/m2 IV bolus on Day 1, q 2wk x4 cycles; 5-FU 2.4g/m2 IV for 46 hours on Day 1, q 2wk x4 cycles; Leucovorin 200mg/m2 IV for 2 hours on Day 1, q 2wk x4 cycles.
  Interventions: Drug: capecitabine; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Radiation: radiation therapy; Drug: Pyridoxine

INTERVENTIONS:
Drug: capecitabine — 825mg/m2 BID, PO, daily
Drug: fluorouracil — Bolus + IV for 46 hrs on Day 1
  Arms: Irinotecan + 5-FU + Leucovorin; Oxaliplatin + 5-FU + Leucovorin
Drug: irinotecan hydrochloride — IV infusion over 90 min on Day 1
  Arms: Irinotecan + 5-FU + Leucovorin; Irinotecan + Oxaliplatin
Drug: leucovorin calcium — 200mg/m2 IV 2 hour infusion on Day 1
  Arms: Irinotecan + 5-FU + Leucovorin; Oxaliplatin + 5-FU + Leucovorin
Drug: oxaliplatin — 85mg/m2 IV infusion for 90minutes on Day 1
  Arms: Irinotecan + Oxaliplatin; Oxaliplatin + 5-FU + Leucovorin
Radiation: radiation therapy — Original Planning Target Volume (PTV1): The total dose to the prescription point shall be 4500 cGy in 25 fractions (Monday - Friday inclusive). Boost Planning Target Volume (PTV2): The cumulative dose within the boost volume to the prescription point shall be 5,040 - 5,400 cGy (per Section 7.5b). Daily Dose: The daily dose to the prescription point of the original and boost volumes shall be 180 cGy. Fractionation: Treatment shall be given 5 days/week. All radiation fields shall be treated once daily.
Drug: Pyridoxine — 50mg TID, PO daily

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, leucovorin, fluorouracil, and oxaliplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well different regimens of induction chemotherapy followed by chemoradiotherapy work in treating patients with locally advanced adenocarcinoma of the rectum.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of obtaining a pre-treatment determination of intratumoral molecular markers (TS, DPD, and ERCC-1) for use in selection of the appropriate regimen for induction cytotoxic combination chemotherapy in patients with cT3-4 rectal adenocarcinoma.
* Determine the response probability (unconfirmed, complete and partial) in patients treated with targeted induction cytotoxic chemotherapy.
* Determine the toxicity of targeted induction cytotoxic chemotherapy and chemoradiotherapy in these patients.
* Determine the response probability in these patients treated with chemoradiotherapy.

OUTLINE: This is a multicenter study.

* Induction chemotherapy: Patients are assigned to 1 of 3 treatment groups based on molecular analysis of the pretreatment tumor specimen.

  * Group I (lower likelihood of resistance to a fluorouracil-based regimen): Patients receive irinotecan IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours beginning on day 1.
  * Group II (higher likelihood of resistance to a fluorouracil-based regimen): Patients receive oxaliplatin IV over 2 hours and irinotecan IV over 90 minutes on day 1.
  * Group III (high likelihood of sensitivity to oxaliplatin and fluorouracil therapy): Patients receive oxaliplatin IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours beginning on day 1.

Treatment in all groups repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are evaluated for response approximately 2 weeks after the completion of induction chemotherapy. Patients with stable disease or better receive chemoradiotherapy.

* Chemoradiotherapy: Beginning approximately 3 weeks after the completion of induction chemotherapy, patients receive oral capecitabine twice daily continuously for 5 weeks and concurrent radiotherapy once daily 5 days a week for 5 weeks.

After chemoradiotherapy, patients may undergo attempted surgical resection at the discretion of the treating physician.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 10-65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary adenocarcinoma of the rectum
* Locally advanced disease (clinical T3-4, N0-2, M0) based on at least 1 of the following criteria:

  * Clinically fixed tumors on rectal examination with tumor adherent to the pelvic sidewall and/or sacrum
  * Sciatica attributed to sacral root invasion with CT scan/MRI evidence of the lack of clear tissue plane is considered evidence of fixation
  * Hydronephrosis on CT scan or intravenous pyelogram of ureteric or bladder invasion by cystoscopy and cytology or biopsy
  * Invasion into the prostate, vagina, or uterus
* Transmural penetration of tumor through the muscularis propria as evidenced by CT scan or MRI and endorectal ultrasound
* Distal border of the tumor must be at or below the peritoneal reflection (within 12 cm of the anal verge) by proctoscopic examination
* Measurable disease by x-ray, scans, or physical examination
* Available tumor tissue to determine molecular profile of the tumor before study treatment
* No clinical evidence of high-grade (lumen diameter < 1 cm) large bowel obstruction unless a diverting colostomy has been performed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,500/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT or SGPT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* See Disease Characteristics
* Creatinine ≤ 1.5 times ULN OR
* Estimated creatinine clearance > 50 mL/min

Cardiovascular

* No significant cardiac disease
* No recent myocardial infarction

Gastrointestinal

* See Disease Characteristics
* Able to swallow oral medication
* No active inflammatory bowel disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No prior unanticipated severe reaction to study drugs
* No known dihydropyrimidine dehydrogenase deficiency
* No serious uncontrolled infection
* No other serious medical illness that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for colon or rectal cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic radiotherapy
* No prior intra-operative radiotherapy or brachytherapy
* No concurrent intra-operative radiotherapy or brachytherapy
* No concurrent intensity-modulated radiotherapy

Surgery

* See Disease Characteristics
* See Radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-08; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Response (confirmed and unconfirmed response, complete response, partial response)

CONTACTS AND LOCATIONS:
Overall Officials: Charles R. Thomas, MD, Study Chair — The University of Texas Health Science Center at San Antonio; Heinz-Josef Lenz, MD, Study Chair — University of Southern California; Robert P. Whitehead, MD, Study Chair — University of Texas; James L. Abbruzzese, MD, Study Chair — M.D. Anderson Cancer Center; Stephen R. Smalley, MD, Study Chair — Radiation Oncology Center of Olathe; Morton S. Kahlenberg, MD, Study Chair — The University of Texas Health Science Center at San Antonio